CLINICAL TRIAL: NCT00329030
Title: Phase III Rituxan/BEAM vs. Bexxar/BEAM With Autologous Hematopoietic Stem Cell Transplantation (ASCT) for Persistent or Relapsed Chemotherapy Sensitive Diffuse Large B-cell Non-Hodgkin's Lymphoma (BMTCTN0401)
Brief Title: Rituxan/BEAM vs Bexxar/BEAM in Autologous Hematopoietic Stem Cell Transplant for Non-Hodgkin's Lymphoma (BMTCTN0401)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0401; BMT CTN 0401 (Other: Blood and Marrow Transplant Clinicial Trials Network); U01HL069294-05 (NIH); 384 (Other: BMT CTN); NCT00415012 (obsolete NCT alias)
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2017-08

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Non-Hodgkin
Keywords: Large B-Cell Lymphoma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Non-Hodgkin | interventions — Rituximab; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituxan/BEAM (Active Comparator): Autologous transplantation using rituxan/BEAM
  Interventions: Drug: Autologous transplantation using rituxan/BEAM
- Bexxar/BEAM (Experimental): Autologous transplantation using Bexxar/BEAM
  Interventions: Drug: Autologous transplantation using Bexxar/BEAM

INTERVENTIONS:
Drug: Autologous transplantation using rituxan/BEAM — Rituxan 375 mg/m2 (Day -19 and Day -12); BCNU 300 mg/m2 (Day -6); Etoposide (VP-16) 100 mg/m2 twice a day (Days -5 to -2); Cytarabine 100 mg/m2 twice a day (Days -5 to -2); Melphalan 140 mg/m2 (Day -1); Followed by autologous transplantation
  Other Names: Rituximab
  Arms: Rituxan/BEAM
Drug: Autologous transplantation using Bexxar/BEAM — Bexxar dosimetric dose 5 mCi (Day -19); Bexxar therapy dose 75 cGy TBD (Day -12); BCNU 300 mg/m2 (Day -6); Etoposide (VP-16) 100 mg/m2 twice a day (Days -5 to -2); Cytarabine 100 mg/m2 twice a day (Days -5 to -2); Melphalan 140 mg/m2 (Day -1); Followed by autologous transplantation
  Other Names: Tositumomab and Iodine I 131 Tositumomab Bexxar
  Arms: Bexxar/BEAM

SUMMARY:
This study is designed as a Phase III, multicenter trial, comparing progression-free survival (PFS) after autologous hematopoietic stem cell transplantation using a standard Rituxan plus BEAM transplant regimen versus a regimen adding Bexxar to BEAM.

DETAILED DESCRIPTION:
BACKGROUND:

Bexxar (Tositumomab and Iodine I 131 Tositumomab) is a radioimmunoconjugate with demonstrated anti-lymphoma effects. This drug is indicated for the treatment of patients with CD20 positive, relapsed or refractory, low grade, follicular, or transformed non-Hodgkin's lymphoma, including patients with Rituximab-refractory non-Hodgkin's lymphoma. Bexxar has been used in several Phase I and II transplant trials either alone or in combination with high-dose chemotherapy for the treatment of relapsed non-Hodgkin's lymphoma. The Phase I and II trials combining Bexxar with BEAM and autologous hematopoietic stem cell transplantation demonstrated promising early results with 80% event-free survival in relapsed chemosensitive diffuse large B-cell non-Hodgkin's lymphoma patients. The administration of Rituxan to the mobilization and conditioning regimen is now the standard of care at most transplant centers. Therefore, the primary endpoint of this study will be to compare progression-free survival after autologous hematopoietic stem cell transplantation for chemotherapy-sensitive diffuse large B-cell lymphoma using Rituxan/BEAM versus Bexxar/BEAM for pre-transplant conditioning.

DESIGN NARRATIVE:

All patients will receive induction or salvage chemotherapy as indicated by their clinical circumstance to achieve at least a partial response (as defined in the protocol). There must be 20% or less bone marrow involvement after their most recent salvage therapy.

Mobilization therapy may be employed per institutional guidelines, but all patients must receive one dose of rituxan (375 mg/m^2) at least within 4 weeks of actual stem cell apheresis. Patients must have an adequate autograft (target of at least 2.0 X 10^6 CD34+ cells/kg; minimum of more than 1.5 X 106 CD34+ cells/kg) to be eligible for the protocol. Eligible patients will be randomized to receive either: 1) Rituxan plus BEAM, with Rituxan 375 mg/m^2 IV Days -19 and -12, Carmustine (BCNU) 300 mg/m^2 Day -6, Etoposide 100 mg/m^2 Days -5 to -2, Cytarabine 100 mg/m^2 Days -5 to -2, and Melphalan 140 mg/m^2 Day -1 followed by ASCT; or, 2) Bexxar/BEAM with the dosimetric dose of 5 mCi Bexxar on Day -19 and the therapeutic dose calculated to administer 75 cGy total body dose (TBD) on Day -12. Patients will then receive BCNU 300 mg/m^2 Day -6, Etoposide 100 mg/m^2 Days -5 to -2, Cytarabine 100 mg/m^2 Days -5 to -2, and Melphalan 140 mg/m^2 Day -1 followed by ASCT.

Patients will be followed for 2 years post-transplant. Survival data, hematopoiesis data, incidence of infection, mucositis assessment data, immune reconstitution data, and toxicity data will be recorded and reported periodically to the BMT CTN Data Coordinating Center (DCC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent or recurrent REAL classification diffuse large B-cell lymphoma, composite lymphoma with more than 50% diffuse large B-cell lymphoma, mediastinal B-cell lymphoma
* Demonstration of CD20+ on at least one histologic specimen
* 18-80 years old at time of first registration
* Three or fewer prior regimens of chemotherapy over the entire course of their disease treatment (including one induction chemotherapy and no more than 2 salvage chemotherapies); monoclonal antibody therapy and involved field radiation therapy will not be counted as prior therapies
* Disease status of primary induction failure, first relapse, or second complete remission; all patients must have chemosensitive disease as demonstrated by response to induction or salvage chemotherapy with at least a partial response (as defined in the protocol)
* No more than a 20% bone marrow involvement
* Patients with adequate organ function as measured by:
* Cardiac: American Heart Association Class I: Patients with cardiac disease but without resulting limitation of physical activity; ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain; additionally, patients greater than 60 years of age must have a left ventricular ejection fraction at rest of at least 40% demonstrated by Multi-Gated Acquisition Scan (MUGA)
* Hepatic: Bilirubin less than 2.0 mg/dL (except for isolated hyperbilirubinemia attributed to Gilbert syndrome) and alanine transaminase (ALT) and aspartate transaminase (AST) less than 3x the upper limit of normal
* Renal: Creatinine less than 2.0 mg/dL or creatinine clearance (calculated creatinine clearance is permitted) more than 40 mL/min; no hydronephrosis on CT scan prior to mobilization
* Pulmonary: Carbon Monoxide Diffusing Capacity (DLCO), Volume forcibly exhaled in one second (FEV1), forced vital capacity (FVC) at least 45% of predicted (corrected for hemoglobin)
* Autologous graft with a minimum of at least 1.5 X 10^6 CD34+ cells/kg (target greater than 2.0 X 10^6 CD34+ cells/kg. Peripheral blood stem cells (PBSC) are preferred; however, if PBSC mobilization fails, cells can be obtained by institutional practices (in cases where bone marrow will be used for transplantation, the required CD34+ dose does not apply and institutional practice for total nucleated cell dose should be used).
* Initiate conditioning therapy within 3 months of mobilization
* Signed informed consent

Exclusion Criteria:

* Karnofsky performance score less than 70%
* Transformed follicular lymphoma
* Uncontrolled bacterial, viral, or fungal infection (currently taking medication and with progression or no clinical improvement)
* Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ; cancer treated with curative intent less than 5 years previously will not be allowed unless approved by the Medical Monitor or Protocol Chair; cancer treated with curative intent less than 5 years previously will be allowed
* Pregnant (positive β-HCG) or breastfeeding; this patient population is excluded due to the lack of data on the use of Bexxar in patients who are pregnant or breastfeeding
* Seropositivity for HIV; this patient population is excluded due to the lack of data on the use of Bexxar in HIV positive patients and because the treatment regimens are too immunosuppressive for this patient population
* Fertile men or women unwilling to use contraceptive techniques from the time of initiation of mobilization until six-months post-transplant
* Prior autologous or allogeneic hematopoietic stem cell transplantation (HSCT)
* Patients with evidence of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML) or abnormal cytogenetic analysis indicative of MDS on the pre-transplant bone marrow examination
* Patients with a prior severe reaction to Rituxan or Filgrastim (G-CSF). Patients with severe reactions to G-CSF that receive pre-medication for control of the reaction are not excluded from study.
* Patients who have received prior radioimmunotherapy
* Patients with known hypersensitivity to murine proteins

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2005-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (36):
- United States (36):
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - St. Lukes Mountain States Tumor Institute, Boise, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Medical Systems/Greenbaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins/SKCCC, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, The New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Columbia River Oncology Program, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - University of Utah Medical School, BMT, Salt Lake City, Utah
  - Intermountain BMT Program, Salt Lake City, Utah
  - Virginia Commonwealth University/MCV Hospital, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Vose JM, Carter S, Burns LJ, Ayala E, Press OW, Moskowitz CH, Stadtmauer EA, Mineshi S, Ambinder R, Fenske T, Horowitz M, Fisher R, Tomblyn M. Phase III randomized study of rituximab/carmustine, etoposide, cytarabine, and melphalan (BEAM) compared with iodine-131 tositumomab/BEAM with autologous hematopoietic cell transplantation for relapsed diffuse large B-cell lymphoma: results from the BMT CTN 0401 trial. J Clin Oncol. 2013 May 1;31(13):1662-8. doi: 10.1200/JCO.2012.45.9453. Epub 2013 Mar 11. PMID 23478060

RESULTS

PARTICIPANT FLOW:
Groups:
- B-BEAM: Patients received Bexxar/BEAM with the dosimetric dose of 5 mCi Bexxar on Day -19 and the therapeutic dose calculated to administer 75 cGy total body dose (TBD) on Day -12. Patients will then receive carmustine (BCNU) 300 mg/m2 Day -6, Etoposide 100 mg/m2 BID Days -5 to -2, Cytarabine 100 mg/m2 BID Days -5 to -2, and Melphalan 140 mg/m2 Day -1 followed by ASCT
- R-BEAM: Patients received Rituxan/BEAM, with Rituxan 375 mg/m2 IV Days -19 and -12, BCNU 300 mg/m2 Day -6, Etoposide 100 mg/m2 BID Days -5 to -2, Cytarabine 100 mg/m2 BID Days -5 to -2, and Melphalan 140 mg/m2 Day -1 followed by ASCT
Period: Overall Study
Arm/Group | B-BEAM | R-BEAM
Started | 111 | 113
Completed | 103 | 107
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Progressive Disease | 6 | 2
Not completed — Ineligible Pathology | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- B-BEAM: Bexxar/BEAM
- R-BEAM: Rituxan/BEAM
- Total: Total of all reporting groups
Arm/Group | B-BEAM | R-BEAM | Total
Number analyzed (Participants) | 111 | 113 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.5) | 56.8 (12.5) | 56.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 68 | 74 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 99 | 101 | 200
  Unknown or Not Reported | 10 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 99 | 103 | 202
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 2 | 6
Primary Disease Stage [Number; unit: participants]
  Primary Induction Failure | 21 | 15 | 36
  First Relapse | 35 | 46 | 81
  Second Complete Remission | 55 | 52 | 107
Karnofsky Performance-status Score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    100% | 29 | 26 | 55
    90% | 67 | 63 | 130
    80% | 12 | 19 | 31
    70% | 3 | 5 | 8
Disease Status at Transplantation [Number; unit: participants]
  First Partial Response | 21 | 15 | 36
  First Relapse | 35 | 45 | 80
  Second Complete Remission | 55 | 53 | 108
Number of Prior Therapies [Number; unit: participants]
  1 | 2 | 7 | 9
  2 | 93 | 83 | 176
  3 | 16 | 23 | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Patients are considered a failure for this endpoint if they die, relapse/progress, or receive anti-lymphoma therapy, other than post-transplant consolidative localized radiation (maximum 3 sites) to sites of prior bulk disease pre-transplant (> 3cm). The time to this event is the time from randomization until death, relapse/progression, receipt of anti-lymphoma therapy, or last follow up, whichever comes first.
Time Frame: 1 and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  1 year | 53.2 [43.5 to 61.9] | 56.6 [46.8 to 65.2]
  2 years | 48.6 [39.0 to 57.5] | 49.0 [39.3 to 58.0]

2. Secondary Outcome: Overall Survival
Description: The event is death from any cause. The time to this event is the time from randomization to death or last follow-up. Surviving patients are censored at the time of last observation
Time Frame: 1 and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  1 year | 68.5 [58.9 to 76.2] | 73.7 [64.4 to 80.9]
  2 years | 60.1 [50.3 to 68.6] | 66.3 [56.6 to 74.3]

3. Secondary Outcome: Incidence of Relapse/Progression
Description: The time to this event is measured from randomization. Deaths without relapse/progression are considered as a competing risk. Surviving patients with no history of relapse/progression are censored at time of last follow-up.
Time Frame: 1 and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  1 year | 39.6 [30.4 to 48.8] | 40.7 [31.5 to 49.9]
  2 years | 44.2 [34.8 to 53.6] | 47.4 [38.0 to 56.8]

4. Secondary Outcome: Complete Response (CR) and Partial Response (PR) Proportion
Time Frame: Day 100 and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  Day 100 | 69.9 [60.1 to 78.6] | 71.0 [61.5 to 79.4]
  2 years | 48.5 [38.6 to 58.6] | 43.9 [34.3 to 53.9]

5. Secondary Outcome: Platelet Recovery to 20,000 Cells/μL
Time Frame: 100 and 180 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  Day 100 | 83.5 [76.2 to 90.8] | 82.2 [74.8 to 89.6]
  Day 180 | 84.5 [77.4 to 91.6] | 83.2 [75.9 to 90.5]

6. Secondary Outcome: Hematologic Function
Description: Hematologic function will be defined as ANC > 1,500 neutrophils/μL, hemoglobin > 10 g/dL without transfusion support, and platelet count > 100,000/μL without transfusion support.
Time Frame: 100 days, 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  Day 100 | 34.8 [25.2 to 45.4] | 38.5 [28.8 to 49.0]
  1 year | 64.0 [52.1 to 74.8] | 58.9 [46.8 to 70.3]

7. Secondary Outcome: Incidence of Infection
Time Frame: 1 year
Population: 67 patients treated with B-BEAM incurred a total of 139 infections. 60 patients treated with R-BEAM incurred a total of 121 infections.
Measure: Number; unit: participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
participants
  1 Infection | 38 | 35
  2 Infections | 14 | 11
  3 Infections | 5 | 7
  4 Infections | 3 | 4
  5 Infections | 1 | 0
  6-10 Infections | 6 | 2
  >10 Infections | 0 | 1

8. Secondary Outcome: Mucositis Severity
Description: Mucositis severity will be scored per the modified Oral Mucositis Assessment Scale (OMAS) scoring system on a scale of 0 - 4, where 0 equals normal mucosa and 4 equals severe mucosa.
Time Frame: Day 21
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
scores on a scale | 0.72 [0.00 to 2.00] | 0.31 [0.00 to 1.75]

9. Secondary Outcome: Immune Reconstitution
Description: Tests to be performed on peripheral blood include CD2, CD3, CD4, CD8, CD19, CD3+/CD25+, CD45 RA/RO, CD56+/CD3-.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
cells/uL
  CD2 (cells/uL) | 1006.0 (767.6) | 1024.9 (1074.7)
  CD3 (cells/uL) | 921.8 (694.8) | 990.3 (1056.1)
  CD4 (cells/uL) | 342.8 (223.9) | 286.1 (213.3)
  CD8 (cells/uL) | 558.5 (517.9) | 697.7 (901.1)
  CD19 (cells/uL) | 143.4 (140.5) | 140.8 (203.0)
  CD3+/CD25+ (cells/uL) | 112.2 (92.8) | 118.0 (127.7)
  CD45RA (cells/uL) | 469.3 (404.4) | 579.8 (620.5)
  CD45RO (cells/uL) | 476.2 (337.4) | 727.8 (798.8)
  CD56+/CD3- (cells/uL) | 125.1 (94.6) | 130.5 (135.7)

10. Secondary Outcome: Immune Reconstitution of Quantitative Immunoglobulins
Description: Tests to be performed on peripheral blood for quantitative immunoglobulins include IgM, IgG and IgA.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
mg/dL
  IgA (mg/dL) | 68.5 (42.6) | 85.0 (71.8)
  IgG (mg/dL) | 619.6 (289.2) | 643.8 (395.3)
  IgM (mg/dL) | 51.0 (36.0) | 79.0 (154.4)

11. Secondary Outcome: Treatment-related Mortality (TRM)
Description: TRM is defined as death occurring in a patient from causes other than relapse or progression
Time Frame: 1 and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  1 year | 5.9 [1.2 to 10.6] | 2.9 [0.0 to 6.0]
  2 years | 5.9 [1.2 to 10.6] | 3.9 [0.2 to 7.6]

12. Secondary Outcome: Neutrophil Recovery
Description: Time to neutrophil recovery will be the first of two consecutive days of > 500 neutrophils/μL following the expected nadir.
Time Frame: Day 28 and Day 60
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B-BEAM | R-BEAM
Number analyzed (Participants) | 103 | 107
percentage of participants
  Day 28 | 96.1 [92.2 to 100.0] | 93.5 [88.6 to 98.4]
  Day 60 | 96.1 [92.2 to 100.0] | 95.3 [91.2 to 99.4]

ADVERSE EVENTS:
Time Frame: Patients will be followed for at least two years post-ASCT.
Description: Serious Adverse Events (AE) are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected grades 3-5 adverse events were required to be reported through the AE system per protocol.
Arm/Group | B-BEAM | R-BEAM
Serious Adverse Events (participants affected / at risk) | 11/111 | 6/113
Other Adverse Events (participants affected / at risk) | 0/111 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-BEAM (N=111) | R-BEAM (N=113)
Acute graft versus host disease in liver (Immune system disorders) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Orchidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Engraft failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-09-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT00329030/Prot_SAP_ICF_000.pdf